CLINICAL TRIAL: NCT06238362
Title: Randomized Crossover Study to Compare Effectiveness of a Device Providing Pressure Drops During Inspiration (TPAP) to Continuous Positive Airway Pressure (CPAP) in Obstructive Sleep Apnea (OSA)
Brief Title: TheraPAP Equivalence Crossover Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SleepRes Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TheraEquivalence
Record Dates: First submitted 2024-01-17; First posted 2024-02-02 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Patients will be treated with both the interventional therapy and standard CPAP therapy in one night to compare efficacy.
Who Masked: Participant
Masking Description: Participants will be asleep during both therapies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- TPAP - Experimental Therapy (Experimental): Experimental therapy in which pressure is reduced during inspiration and the reduction is carried through part of expiration such that the pressure is increased near the end of expiration.
  Interventions: Other: TPAP
- CPAP - Traditional OSA Therapy (Active Comparator): Standard OSA therapy to which the TPAP therapy will be compared for efficacy.
  Interventions: Device: CPAP

INTERVENTIONS:
Other: TPAP — Algorithm for modification of CPAP therapy where pressure is reduced during the inspiratory phase though much of the expiratory phase, then is returned to full pressure near the end of the expiratory phase. Note that the same device that delivers CPAP can also deliver TPAP
  Other Names: TheraPAP
  Arms: TPAP - Experimental Therapy
Device: CPAP — Gold standard for treating sleep apnea.
  Arms: CPAP - Traditional OSA Therapy

SUMMARY:
The present study, TheraEquivalence, is a Phase 2 crossover study designed to examine the efficacy and safety of TheraPAP (TPAP) vs. CPAP alone in the treatment of OSA.

DETAILED DESCRIPTION:
The TheraEquivalence Study is a randomized, controlled, crossover study in participants with OSA. A split-night polysomnogram (PSG) will be conducted on CPAP and TPAP (3.5 h each treatment arm) in previously diagnosed OSA patients, to test the effectiveness of TPAP vs. CPAP. The sequence of periods for each participant are assigned in random order. Therapeutic CPAP level will be defined based on each individual's pressure levels from their currently used APAP device deemed to eliminate breathing obstructions for at least 90/95% of the sleep period (P90/P95) + 1 cmH2O (cm of water pressure). P90/P95 will be defined based on the previous 2 months of adherent Auto-adjusted Positive Airway Pressure (APAP) usage (defined as averaging > 5 hrs/night). On TPAP Tthe pressure drop during inspiration is generally done in two steps and varies, as outlined in table 1, based on the set pressure level, with larger drops occurring when the set pressure is higher. However, the pressure never goes below 5 cm H20. This lower pressure is returned to the set pressure level about halfway through expiration. These pressure drops are designed to make TPAP considerably more comfortable than CPAP.

ELIGIBILITY:
Inclusion Criteria:

1. AHI > 10 on a previous PSG.
2. CPAP adherence for an average of 5 h/night in the 2 months before the study
3. BMI above 18 kg/m2, inclusive.

Exclusion Criteria:

1. Current clinically significant sleep disorder other than OSA of a severity that would interfere with study participation or interpretability of data (including central sleep apnea, per central AHI > 5 events/h).
2. Current clinically unstable cardiac disease (e.g., rhythm disturbances, coronary artery disease or cardiac failure) or poorly controlled hypertension (>140/90mmHg).
3. Current clinically significant neurological disorder, including epilepsy/convulsions.
4. Other serious major organ system disease including renal failure, lung disease, neuromuscular disease, or liver disease.
5. Schizophrenia, schizoaffective disorder or bipolar disorder according to Diagnostic and Statistical Manual of Mental Disorders-5 (DSM 5) or International Classification of Disease tenth edition criteria.
6. Attempted suicide within 1 year prior to screening, or current suicidal ideation.
7. History of substance use disorder as defined in DSM-V within 24 months prior to Screening Visit.
8. A serious illness or infection in the past 30 days as determined by investigator.
9. Clinically significant cognitive dysfunction as determined by investigator.
10. Chronic oxygen therapy.
11. Patients with hypoglossal nerve stimulation implant.
12. Any non-previously mentioned vulnerable population.
13. Any condition that in the investigator's opinion would present an unreasonable risk to the participant, or which would interfere with their participation in the study or confound study interpretation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abinash Joshi, MD, Principal Investigator — SleepRes Inc.
Locations (1):
- SleepCenters of Middle Tennessee, Clarksville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: CPAP First TPAP Second; Sequence 2: TPAP First CPAP Second: CPAP first: set on P90/P95+1cmH2O TPAP second: two drops of maximum 5cmH2O starting from baseline pressure, one at the start of inspiration, the other at peak inspiratory flow
Period: Overall Study
Arm/Group | Sequence 1: CPAP First TPAP Second | Sequence 2: TPAP First CPAP Second
Started | 28 | 22
Completed | 26 | 22
Not Completed | 2 | 0
Not completed — Insufficient total sleep time | 1 | 0
Not completed — Inadequate signal quality | 1 | 0

BASELINE CHARACTERISTICS:
Population: This number includes 2 people who were excluded from the final analysis
Groups:
- Overall Group: The study was a crossover trial of two treatment administered over the same night.
Arm/Group | Overall Group
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 43
  More than one race | 0
  Unknown or Not Reported | 0
P90/P95 [Mean (Standard Deviation); unit: cmH2O] — P90/P95 is the positive pressure delivered by the device for 90 or 95% of the night, respectively
  cmH2O | 10.6 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Apnea/Hypopnea Index
Description: Gold standard measure of CPAP therapy efficacy. Scored as number of respiratory events per hour of sleep. The device is considered efficacious with an apnea-hypopnea index < 5 events/h.
Time Frame: During overnight procedure, on average 3.5 hours for each intervention
Measure: Mean (Standard Deviation); unit: events/h
Arm/Group | TPAP - Experimental Therapy | CPAP - Traditional OSA Therapy
Number analyzed (Participants) | 48 | 48
events/h | 2.9 (4.1) | 3.2 (3.9)

2. Secondary Outcome: REM Apnea/Hypopnea Index (AHI)
Description: Scored as number of respiratory events per hour of sleep spent in rapid eye movement stage. The device is generally considered efficacious with an apnea-hypopnea index in REM < 5 events/h, however it has to be noted that obstructive sleep apnea during REM sleep is more difficult to treat.
Time Frame: During rapid eye movements (REM) sleep during the overnight procedure, assessed over 3.5 hours for each intervention
Population: Some people did not have REM sleep, hence the reduced participant sample
Measure: Mean (Standard Deviation); unit: events/h
Arm/Group | TPAP - Experimental Therapy | CPAP - Traditional OSA Therapy
Number analyzed (Participants) | 43 | 43
events/h | 4.3 (5.1) | 6 (6.8)

3. Secondary Outcome: Supine AHI
Description: Assessment of AHI (apnea hypopnea index) during supine sleep. The device is generally considered efficacious if supine AHI is below 5 events/h, however it has to be noted that obstructive sleep apnea in supine position is more difficult to treat.
Time Frame: During sleep spent in supine position during the overnight procedure, assessed over 3.5 hours for each intervention
Population: Some people did not sleep in supine position, thus the participant sample is reduced
Measure: Mean (Standard Deviation); unit: events/h
Arm/Group | TPAP - Experimental Therapy | CPAP - Traditional OSA Therapy
Number analyzed (Participants) | 40 | 40
events/h | 4.9 (7.5) | 5.4 (6.9)

4. Secondary Outcome: Unintentional Patient Circuit Leak
Description: Evaluation of unintentional circuit leak by measuring flow offset from CPAP and knowing the intentional mask leak
Time Frame: During overnight procedure
Population: With some machine, it was not possible to determine the leak with precision, hence the reduced participant sample
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | TPAP - Experimental Therapy | CPAP - Traditional OSA Therapy
Number analyzed (Participants) | 45 | 45
L/min | 2.8 (3.6) | 5.1 (4.3)

5. Secondary Outcome: NREM Apnea/Hypopnea Index (AHI)
Description: Scored as number of respiratory events per hour of sleep spent in non-rapid eye movement stage (NREM). The device is generally considered efficacious with an apnea-hypopnea index in NREM < 5 events/h.
Time Frame: During non-rapid eye movements (NREM) sleep during the overnight procedure, assessed over 3.5 hours for each intervention
Measure: Mean (Standard Deviation); unit: events/h
Arm/Group | TPAP - Experimental Therapy | CPAP - Traditional OSA Therapy
Number analyzed (Participants) | 48 | 48
events/h | 2.3 (4.4) | 2.2 (3.7)

6. Secondary Outcome: Lateral AHI
Description: Assessment of AHI (apnea hypopnea index) during lateral sleep. The device is generally considered efficacious if lateral AHI is below 5 events/h
Time Frame: During sleep spent in lateral position during the overnight procedure, assessed over 3.5 hours for each intervention
Population: Some people did not sleep in lateral position, thus the participant sample is reduced
Measure: Mean (Standard Deviation); unit: events/h
Arm/Group | TPAP - Experimental Therapy | CPAP - Traditional OSA Therapy
Number analyzed (Participants) | 39 | 37
events/h | 2.4 (5.4) | 3 (5.8)

ADVERSE EVENTS:
Time Frame: 1 night (half night for each treatment)
Arm/Group | TPAP - Experimental Therapy | CPAP - Traditional OSA Therapy
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 1/50 | 0/50
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPAP - Experimental Therapy (N=50) | CPAP - Traditional OSA Therapy (N=50)
Insufficient sleep (Nervous system disorders) | 1 (1) | 0 (0) — The participant did not get a sufficient sleep time on the treatment arm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT06238362/Prot_SAP_001.pdf